CLINICAL TRIAL: NCT07274917
Title: The Efficacy and Safety of Stereotactic Radiotherapy for Treatment-Resistant Depression: An Open-Label Exploratory Study
Brief Title: Stereotactic Radiotherapy Treatment for Treatment-resistant Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, Dean of Beijing Anding Hospital, Capital Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025(60)
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Treatment-Resistant Depression; Depressive Disorder
Keywords: Treatment-Resistant depression; X-ray; subgenual anterior cingulate cortex; ZAP-X; stereotactic radiotherapy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Intervention Group: 15Gy (Experimental): All patients will then undergo 3 (minimum)-7 (maximum) MRI scans during baseline preparation period, with intervals of more than 24 hours between scans. Based on the axial 3D-T1 weighted image, the anterior commissure (AC) and posterior commissure (PC) are determined. Select the sagittal T2 image and identify the cingulate sulcus below the genu of the corpus callosum. Draw a line from the genu of the corpus callosum to the anterior commissure and take the midpoint. Then, on the coronal T2 image, locate the coronal section corresponding to this midpoint as the target point.
  The treatment schedule was as follows: each patient received unilateral irradiation per day at a dose of 15 Gy, with each session lasting approximately 20 minutes. The entire treatment was completed over two days, and the isodose lines were set at 80%
  Interventions: Device: ZAP-X
- Intervention Group: 20Gy (Experimental): All patients will then undergo 3 (minimum)-7 (maximum) MRI scans during baseline preparation period, with intervals of more than 24 hours between scans. Based on the axial 3D-T1 weighted image, the anterior commissure (AC) and posterior commissure (PC) are determined. Select the sagittal T2 image and identify the cingulate sulcus below the genu of the corpus callosum. Draw a line from the genu of the corpus callosum to the anterior commissure and take the midpoint. Then, on the coronal T2 image, locate the coronal section corresponding to this midpoint as the target point. The treatment schedule was as follows: each patient received unilateral irradiation per day at a dose of 20Gy, with each session lasting approximately 20 minutes. The entire treatment was completed over two days, and the isodose lines were set at 80%
  Interventions: Device: ZAP-X
- Intervention Group: 25 Gy (Experimental): All patients will then undergo 3 (minimum)-7 (maximum) MRI scans during baseline preparation period, with intervals of more than 24 hours between scans. Based on the axial 3D-T1 weighted image, the anterior commissure (AC) and posterior commissure (PC) are determined. Select the sagittal T2 image and identify the cingulate sulcus below the genu of the corpus callosum. Draw a line from the genu of the corpus callosum to the anterior commissure and take the midpoint. Then, on the coronal T2 image, locate the coronal section corresponding to this midpoint as the target point. The treatment schedule was as follows: each patient received unilateral irradiation per day at a dose of 25 Gy, with each session lasting approximately 20 minutes. The entire treatment was completed over two days, and the isodose lines were set at 80%
  Interventions: Device: ZAP-X

INTERVENTIONS:
Device: ZAP-X — The individualized bilateral sgACC template will be imported into the ZAP-X treatment planning system. For left and right sgACC targets, the treatment plan will be automatically generated with the following set-up. The treatment will be carried out on two consecutive days.

SUMMARY:
This study is an clinical trial aimed at evaluating the effectiveness and safety of stereotactic radiotherapy for treatment-resistant depression

DETAILED DESCRIPTION:
Treatment-Resistant Depression (TRD) generally refers to patients with depression who have received at least two antidepressants with different mechanisms of action, at adequate doses and for sufficient durations, but have shown poor or no response. TRD is difficult to treat and usually has a poor prognosis, seriously affecting the normal life of patients and their families. One of the imaging manifestations of TRD patients is abnormal functional activity of the subgenual anterior cingulate cortex (sgACC). The direct clinical intervention method for this area is to implant a deep brain stimulator through an invasive approach. However, this intervention method has a low risk-benefit ratio and is poorly accepted by patients.

Radiation is a widely used clinical intervention technique. By focusing rays from multiple angles, it can generate high-energy rays in a local area of the human brain for ablation. This technique is typically used for targeted ablation of tumors and has the advantage of high precision. Recently, breakthrough research has found that radiotherapy can be applied in the field of psychiatry. In experiments with doses of 10Gy and 20Gy, researchers observed an increase in the standard uptake value of the irradiated target area compared to the contralateral brain region in PET images of the subjects, suggesting that radiotherapy can up-regulate glucose metabolism levels without killing neurons at low doses. These clinical studies suggest that stereotactic radiotherapy can safely regulate brain function. Based on this, this project aims to explore the safety, efficacy, and biological mechanisms of low-dose radiotherapy targeting the sgACC in the treatment of TRD.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients or inpatients aged 18 to 50 years (inclusive), regardless of gender.
* Meet the diagnostic criteria for Major Depressive Disorder (MDD), recurrent, without psychotic features, as defined by The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* Documented treatment-resistant depression, defined as a lack of clinically meaningful response (less than 50% improvement in depressive symptoms) to at least two adequate antidepressant trials during the current episode, as recorded by the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (MGH-ATRQ). An adequate trial requires sufficient dosage (within the recommended therapeutic range) and duration (at least 6 weeks). The current episode must involve at least one treatment failure.
* A Hamilton Depression Rating Scale 17-item (HAMD-17) total score of ≥ 20 at both the screening and baseline visits.
* The subject agrees to maintain their existing baseline antidepressant therapy regimen unchanged throughout the study period.
* The patient and their legal guardian understand and voluntarily agree to participate in this study, are capable of adhering to the treatment protocol, and provide written informed consent.

Exclusion Criteria:

* A current or prior diagnosis of any other DSM-5 mental disorder, including but not limited to: neurodevelopmental disorders, bipolar and related disorders, obsessive-compulsive and related disorders, schizophrenia spectrum and other psychotic disorders, substance-related and addictive disorders, or personality disorders.
* A past medical history or current presence of clinically significant somatic diseases, such as severe or unstable cardiovascular, respiratory, digestive, endocrine, urinary, hematological, or nervous system diseases, or benign/malignant tumors; or any condition deemed by the investigator to pose a potential risk to patient safety or their ability to fully participate in the study.
* Any severe neurological disease or impairment, including but not limited to: any condition potentially associated with increased intracranial pressure, space-occupying brain lesions, cerebral infarction, intracranial hemorrhage, history of epileptic seizures or family history of epilepsy (except for those induced by ECT), cerebral aneurysm, Parkinson's disease, Huntington's disease, multiple sclerosis, or a history of severe head trauma with loss of consciousness; or any condition deemed by the investigator to pose a potential risk to patient safety or their ability to fully participate in the study.
* Assessed by the investigator as being at significant risk of suicide, evidenced by: a "Yes" response to Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) in the "Suicidal Ideation" section of the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past 6 months; OR a "Yes" response to any item in the "Suicidal Behavior" section of the C-SSRS (actual attempt, interrupted attempt, aborted attempt, preparatory acts or behavior) within the past 6 months; OR a score of ≥5 on Item 10 (Suicidal Thoughts) of the Montgomery-Åsberg Depression Rating Scale (MADRS).
* Participation in other systematic neuromodulation therapies (e.g., MECT, rTMS, tDCS, VNS, DBS) within 3 months prior to screening, or participation in an interventional clinical trial within 1 month prior to screening.
* Patients who have been non-responsive to a systematic course of MECT treatment.
* Patients with a history of other psychosurgical procedures (including radiofrequency ablation, focused ultrasound, etc.).
* A history of prior radiotherapy, chemotherapy, or immunotherapy, or a history of occupational exposure to radiation/toxic substances.
* Contraindications to Magnetic Resonance Imaging (MRI), including but not limited to: intracranial or bodily metallic implants, implanted pacemakers or cochlear implants, or claustrophobia.
* Pregnant or lactating women.
* Subjects of either gender who plan to become pregnant within the next 6 months or are unwilling to use effective contraception.
* Subjects with a body weight exceeding 150 kg.
* Any other condition considered by the investigator to make the subject unsuitable for participation in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Montgomery-Åsberg Depression Rating Scale (MADRS) score at 4 weeks post-treatment compared to baseline | Pre-treatment and 4 weeks post treatment
  A ten item questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.

SECONDARY OUTCOMES:
Change in the Montgomery Asberg Depression Rating Scale (MADRS) | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  A ten item diagnostic questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.
Change in Columbia Suicide Severity Rating Scale (C-SSRS) score post-treatment | Pre-treatment to post-treatment(week 1, week2, week4, week8, week12)
  A suicidal ideation rating scale created by researchers at Columbia University. The score was calculated by summing the answers to 5 questions. Score range - 0 to 5. Higher score indicate higher suicidal ideation.
Change in Quick Inventory of Depressive Symptomatology (QIDS-SR-16) score post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week 8, week12)
  The QIDS-SR16 consists of 16 items, with each item ranging between 0 and 3 points. The total score ranged from 0 to 27 with higher score implicated severe depressive symptoms.
Change in clinical global impression-severity(CGI-S) post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  The Clinical Global Impression - Severity (CGI-S) is a single-item, clinician-rated scale used to assess the overall severity of a patient's illness. The rating is based on the clinician's total experience with this patient population. It is scored on a 7-point scale, ranging from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients), with higher scores indicating greater illness severity.
Change in clinical global impression-improvement(CGI-I) post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  The Clinical Global Impression - Improvement (CGI-I) is a single-item, clinician-rated scale used to assess how much a patient's illness has improved or worsened since the start of treatment. It is scored on a 7-point scale, ranging from 1 (Very much improved) to 7 (Very much worse), with a score of 4 representing "No change". The rating is based on the clinician's assessment of the patient's overall clinical state.
Change in Instant Mood Scale-12 post-treatment | Pre-treatment to immediate during treatment(on day 1, day 2) and post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  The Instant Mood Scale-12 (IMS-12) is a brief, 12-item self-report questionnaire designed to rapidly assess the current severity of depression and anxiety symptoms.Each item is rated on a 7-point Likert scale (0="Not at all" to 7="Extremely") based on the patient's feelings at the present moment. Total scores for each subscale range from 0 to 84, with higher scores indicating greater symptom severity.
Change in Hamilton Anxiety Scale(HAMA) post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  A 14-item, clinician-administered scale designed to assess the severity of a patient's anxiety. Scores range from 0-56, with higher scores reflecting greater anxiety severity.
Change in Digital Span Test score post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  A test of working memory and attention where participants repeat sequences of auditorily presented numbers, both in forward and backward order. The primary outcome is the longest sequence correctly recalled.
Change in Digit Symbol Substitution Test post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  The Digit Symbol Substitution Test (DSST) is a performance-based neuropsychological test that assesses processing speed, sustained attention, and visual-motor coordination. The test presents the participant with a key pairing nine numbers (1-9) with nine unique symbols. The main task requires the participant to fill in blank spaces with the corresponding symbol for a series of randomly ordered numbers as quickly and accurately as possible within 90 seconds. The primary score is the total number of correct symbol substitutions completed within the time allowed.
Change in Perceived Deficits Questionnaire - Depression score post-treatment | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  The Perceived Deficits Questionnaire - Depression (PDQ-D) is a 20-item self-report scale designed to measure a patient's subjective experience of cognitive dysfunction. It assesses perceived difficulties in four key cognitive domains: attention/concentration (5 items), retrospective memory (5 items), prospective memory (5 items), and planning/organization (5 items). Patients rate the frequency of these cognitive problems over the past week on a 5-point scale from 0 ("Never") to 4 ("Almost always"). A total score is calculated (range 0-80), with higher scores indicating greater perceived cognitive deficits.

OTHER OUTCOMES:
Neuroimaging markers at 4/12 week post-treatment compared to baseline | 4/12 week post-treatment
Electroencephalographic (EEG) markers at 4/12week post-treatment compared to baseline | 4/12 week post-treatment
Digital phenotype post-treatment compared to baseline | Pre-treatment to post-treatment(on day 3, week 1, week 2, week 4, week8, week12)
  Including Audio and video

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Medical Doctor, Principal Investigator — Beijing Anding Hospital, Capital Medical University; Longsheng Pan, Medical Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Beijing Anding Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided